CLINICAL TRIAL: NCT07028983
Title: Fighting Addictions, Improving Lives Through COmprehensive Drug Rehabilitation With Music (FALCO): International Randomised Controlled Trial
Brief Title: Fighting Addictions, Improving Lives: COmprehensive Drug Rehabilitation With Music
Acronym: FALCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: University of Bergen (Other); Helse Stavanger HF (Other Government); Sykehuset Innlandet HF (Other); University of Vienna (Other); Anton Proksch Institut (Unknown); University of Music and Performing Arts, Vienna (Unknown); Austrian Institute for Health Technology Assessment GmbH (Unknown); Herzog College (Unknown); Bar-Ilan University, Israel (Other); University of Pavia (Other); University of Gdańsk (Unknown); Wojewódzki Ośrodek Terapii Uzależnień w Gdańsku (Unknown); Institut d'Investigació Biomèdica de Bellvitge (Other); Institució Catalana de Recerca i Estudis Avançats (Unknown); Universitat de Girona (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Fundació Sanitària d'Igualada (Unknown); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107278; 101155881 (Other Grant/Funding Number: Horizon Europe); REF-1131-52304 (Other Grant/Funding Number: SERI)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: substance use disorder; addiction; recovery; music therapy; mental health; brain health
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary outcome and all other clinician-based measures will be conducted by masked assessors. Masking success will be verified by asking the assessor at the end of the primary endpoint assessment if they inadvertently found out the participant's allocation, and if so, to state the condition they believe the participant was allocated to. Statisticians conducting analyses will also be masked, and report writing will be masked until a draft is ready.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Music Group(AMG) + Treatment as Usual(TAU) (Experimental): Participants will partake in an active music group, as well as undergo treatment as usual as offered locally.
  Interventions: Behavioral: Active Music Group (AMG)
- Music Listening Group(MLG) + Treatment as Usual(TAU) (Experimental): Participants will partake in a music listening group, as well as undergo treatment as usual as offered locally.
  Interventions: Behavioral: Music Listening Group (MLG)
- Treatment as Usual (TAU) (Active Comparator): Treatment as usual, as offered locally and not facilitated by the study.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Active Music Group (AMG) — Active music group is a music therapy intervention where participants actively make/play music in groups. The sessions will be conducted by an appropriately qualified music therapist.
  Arms: Active Music Group(AMG) + Treatment as Usual(TAU)
Behavioral: Music Listening Group (MLG) — Music listening group is a music therapy intervention where participants partake in music listening in groups. The sessions will be conducted by an appropriately qualified music therapist.
  Arms: Music Listening Group(MLG) + Treatment as Usual(TAU)
Behavioral: Treatment as Usual (TAU) — Treatment as usual as provided locally, which may include pharmacological and/or non-pharmacological interventions (e.g. mindfulness-based intervention, structured physical activity).
  Arms: Treatment as Usual (TAU)

SUMMARY:
FALCO is a parallel pragmatic randomized control trial addressing long-term effects of music therapy (MT) on substance use disorder (SUD).

600 participants will be recruited from 7 countries (Norway, Austria, Israel, Italy, Poland, Spain, Switzerland), involving 10 recruitment sites. They will be randomized into one of the following intervention arms: Active Music Group (AMG), Music Listening Group (MLG) or Treatment as Usual (TAU) as offered locally.

DETAILED DESCRIPTION:
Substance use disorder (SUD) is associated with a high global burden of disease: 4.2% of all disability-adjusted life years lost (DALYs, a combined measure of years of life lost and years lived with disability) are due to alcohol and 1.3% due to illicit drugs. Remarkably, approved pharmacological treatment options are not available for most SUDs, and non-pharmacological approaches are still the backbone of SUD treatment.

Music therapy (MT) is a non-pharmacological intervention recommended i some SUD guidelines. In MT, defined as the clinical and evidence-based use of music interventions to accomplish individualized goals within a therapeutic relationship by a credentialed professional, a music therapist uses music and musical activities to support individuals or groups in reaching specific therapeutic goals. This includes activities such as music listening and active music making, which are tailored to participants' cultural context and individual needs.

The FALCO-trial is a parallel 3-arm assessor- and statistician-blinded pragmatic multinational randomized clinical trial. The interventions of interest in the trial (AMG, MLG) are non-pharmacological psychosocial interventions. Both AMG and MLG will be conducted by appropriately qualified music therapists, in groups, with weekly sessions lasting up to 90 minutes. Participants will continue to receive TAU as offered locally.

The primary objective of the study is to determine effects of AMG and MLG versus TAU on addiction severity in people with SUD at one year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* patients seeking or receiving treatment at the recruitment site for an existing substance use disorder based on ICD-10 criteria
* ≥18 years old
* not currently undergoing detoxification (detoxification has been completed or is not currently planned at the time of recruitment)
* any type of substance use including polysubstance and alcohol use

Exclusion Criteria:

* exclusively nicotine dependence
* psychotic episode in the last 3 months
* insufficient language skills to participate in treatment without the use of a translator
* hearing impairment that considerably impairs hearing of music played at a moderate volume (not relevant if hearing is sufficiently compensated by a hearing aid)
* existing diagnosis of dementia
* is currently receiving music therapy or has received music therapy (i.e. at planned and reoccurring intervals, not counting single random occurrences) during the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2037-06-30 (Estimated)

PRIMARY OUTCOMES:
Addiction Severity assessed by the the European Addiction Severity Index (EuropASI) | Baseline, 1 year, 2 years.
  The survey covers a broad concept of addiction, including changes that typically require a long time, across seven domains (general medical condition, professional and financial situation, substance use, other drug consumption, legal problems, family and social relations, psychological condition).
  It has been adapted specifically for use in European contexts. The scale is clinician-based and includes 164 items, with a fine-grained Composite score of 0 (best) to 1 (worst).

SECONDARY OUTCOMES:
Recovery assessed by the Substance Use Recovery Evaluator (SURE) | Baseline, 1 year, 2 years.
  The scale captures five factors (substance use, material resources, outlook on life, self-care, relationships) using 21 items. Each question scores between 1-3. Total score ranges between 21-63, with a higher score indicating better recovery.
  The scale is patient-reported and was developed with strong user involvement.
Substance use severity assessed by Drug Disorder Identification Test (DUDIT-C) | Baseline, 3 months, 1 year, 2 years.
  This scale is a patient-reported short screening tool that can be used repeatedly. It consists of 11 questions, including 9 ranging from 0-4 and 2 from 0-2, producing a DUDIT sum score of 0-40. In addition, a DUDIT-C sum score of the first 4 items can range from 0-16. Higher scores indicate higher substance use severity. A score of 0 indicates self-reported abstinence, scores ≥ 7 indicate heavy use.
Substance use severity assessed by Alcohol Use Disorder Identification Test (AUDIT-C) | Baseline, 3 months, 1 year, 2 years.
  This scale is a patient-reported short screening tool that can be used repeatedly. It consists of 10 questions, each ranging from 0-4, producing an AUDIT sum score of 0-40. In addition, an AUDIT-C sum score of the first 3 items can range from 0-12. Higher scores indicate higher substance use severity. A score of 0 indicates self-reported alcohol abstinence, scores ≥ 3/4 (women/men) indicate alcohol misuse.
Quality of life assessed by EuroQol (EQ-5D) | Baseline, 1 year, 2 years.
  EQ-5D is a patient-reported scale with 5 items plus a visual analogue scale (VAS).
  The 5-item scale ranges from "less than 0" (worse than death; depending on country-specific weights) to 1 (best). The VAS provides a global one-item rating of current perceived health ranging from 0 (worst possible) to 100 (best possible health).
Depressive symptoms assessed by the Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, 1 year, 2 years.
  MADRS is a clinician-administered ten-item interview measuring symptoms of depression. The scale assesses severity of depressive symptoms (rating symptoms on a 7-point scale). Scores range from 0-6, with a maximum score of 60. A higher score indicates more severe depression.
Attrition assessed by clinicians | 3 Months, 1 year, 2 years.
  Clinicians will judge whether a participant is still participating, has decided to withdraw from the study, or contact has been lost. Importantly, participants will not be regarded as withdrawn if they decide to withdraw from interventions or from some assessment procedures.
Adverse effects assessed by clinicians | 3 months, 1 year, 2 years.
  We will ask participants to describe any adverse events, and clinicians will then rate whether these were serious or non-serious and related or non-related.
Employment monitored by public records | 10 years.
  Patients' participation in the study ends after two years. From public records that are unaffected by loss of contact, employment will be monitored until 10 years after randomisation.
Hospitalisation monitored by health records | 10 years.
  Patients' participation in the study ends after two years. From electronic health records unaffected by loss of contact, hospitalisation will be monitored until 10 years after randomisation.
Criminal record monitored by public records | 10 years.
  Patients' participation in the study ends after two years. From public records that are unaffected by loss of contact, criminal record will be monitored until 10 years after randomisation.
Survival monitored by public records | 10 years.
  Patients' participation in the study ends after two years. From public records that are unaffected by loss of contact, survival will be monitored until 10 years after randomisation.
Motivation for change assessed by the Importance, Confidence, Readiness Ruler (ICR) | 1 week, 3 months, 1 year.
  The ICR is a patient-reported scale that assesses overall motivation to change, including readiness to change. It has 3 items and is rated on a 10-point Likert scale, and total scores range from 0 to 30. Higher scores indicate higher motivation to change.
Craving assessed by the Craving Scale | Baseline, 1week, 3 months, 1 year.
  The Craving Scale is a 3-item patient-reported scale. Scores range from 0-9. High scores indicate higher cravings.
Social connectedness assessed by the Inclusion of Other in the Self Scale (IOS) | 1 week, 3 months, 1 year.
  The IOS is a patient-reported single-item visual scale of closeness. scores range from 1-7, with higher score indicating higher social connectedness.
Motivation for change assessed by the University of Rhode Island Change Assessment (URICA) | Baseline, 3 months, 1 year.
  A more comprehensive patient-reported scale than the brief ICR mentioned above. URICA has 32 items and measures the extent to which individuals identify with different stages of change (precontemplation, contemplation, action, maintenance). Each subscale consists of eight items using 5-point Likert scales ranging from 1 to 5 (resulting in scores ranging from 8 to 40). Subscale scores can be used to trace changes in attitudes related to the specific stages of change. The subscales are combined arithmetically (Contemplation + Action + Maintenance - Precontemplation) to yield a Readiness to Change score, with a possible range of 16-80 and higher scores indicating greater readiness for change.
Anhedonia assessed by the Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, 3 months, 1 year.
  SHAPS is a patient-reported scale with 14 items. It measures the capacity to derive pleasure from four different hedonic experiences: interest/pastimes, social interaction, sensory experience and food/drink. Scores range from 0-4. Higher scores represent higher anhedonia level and a lower hedonic tone.
Sleep quality assessed by the Sleep Condition Indicator (SCI) | Baseline, 3 months, 1 year.
  The SCI has 8 questions covering various sleep aspects such as: sleep onset delay, night-time awakenings, extent of the problem and its effect on daytime activities, mood and relations. Responses are scored from 0 (poor state) to 4 (no/minor problems). A total score of ≤ 16 indicates probable insomnia. Maxmimum score is 32.
Substance use measured by hair samples | Baseline, 3 months, 1 year.
  Objective measures of substance use will be assessed through hair testing. Three strands of hair as thick as a matchstick will be collected from the occiput as close to the scalp as possible. The 3 cm most proximal to the scalp will be analysed. The levels of substance use will be quantitatively determined by liquid chromatography-tandem mass spectrometry (LC-MS/MS) using a protocol deriving the maximum amount of high-quality valid information from the smallest amount of hair.
Brain pathology measured from blood samples | Baseline, 3 months, 1 year.
  Neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP) will be used as potential functional biomarkers of individual substance use burden of the brain. NfL and GFAP analysis: Serum will be collected in silica tubes. After 30min clotting time, the samples will be centrifuged with 1500g for 15min at room temperature. Storage temperature will be -80°C. NfL and GFAP concentrations will be measured in triplicates using simple-plex assays (ProteinSimple, CA, USA) on Ella microfluidic system (BioTechne, MN, USA).
Cognitive function assessed by four tests from the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 1 year.
  The selected CANTAB tasks:
  1. Rapid Visual Information Processing (RVP):
     This task focuses on sustained attention.
  2. Spatial Working Memory (SWM):
     This task mainly assesses visuospatial working memory.
  3. Paired Associates Learning (PAL):
     This task measures visuospatial declarative learning and memory.
  4. Intra-Dimensional/Extra-Dimensional Set-Shifting (ID/ED):
  This test covers rule acquisition and reversal, featuring visual discrimination and attentional set-shifting analogous to the Wisconsin Card Sorting Task.
Social cognition assessed by the video-based online test COgnition of Social Interaction in MOvies (COSIMO) | Baseline, 3 months, 1 year.
  COSIMO will measure cognitive empathy and mental perspective taking. Performance will be assessed as number of correct answers.
Creativity assessed by a shortened version of the Test of Creative Imagery Abilities (TCIA) | Baseline, 3 months, 1 year.
  The shortened version of TCIA will be used to measure creative imagery abilities. Participants will be asked to view simple graphite images, generate transformation ideas and draw their favorite idea on paper with no time limit, with the possibility of elaborating or changing the selected image. They will also be asked to write what their drawing represents.
  The level of creative imagery will be measured by scoring the drawings according to three characteristics: vividness, originality, and transformative ability.
Structural brain scans indicating cognitive impairment | Baseline, 3 months, 1 year.
  1. Morphometric analysis (MRI-Voxel Based Morphometry, VBM):
     This analysis permits statistical estimation of whole-brain voxel-level local changes in volume.
  2. Cortical folding and cortical thickness:
     Geometrical representations for the cortical surfaces of each patient will be reconstructed and compared based on 3d/T1-images.
  3. Diffusion Tensor Imaging (MRI-DTI) analysis:
     DTI will provide precise indices related to tissue white-matter integrity and microstructure reorganization.
  4. DRI fiber tracking:
  Tracking and reconstruction of white-matter tracks allow to study the larger scale patterns of connectivity and differences in the major association paths in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gold, PhD, Principal Investigator — NORCE Research Centre
Locations (11):
- Anton Proksch Institut, Vienna, Austria
- Herzog College, Jerusalem, Israel
- University of Pavia, Pavia, Italy
- Norway (3):
  - University of Bergen / NORCE Research AS, Bergen
  - Sykehuset Innlandet, Innlandet
  - Stavanger Universitetssjukehus, Stavanger
- Palestine National Rehabilitation Centre, Bethlehem, Palestinian Territories
- WOTU / University of Gdansk, Gdansk, Poland
- Spain (2):
  - Fundacio Sanitaria d'Igualada, Barcelona
  - IDIBGI, Girona
- CAD, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified curated data will be made available permanently in publicly accessible repositories (e.g. OSF.io) using FAIR principles (e.g. using digital object identifiers [DOIs]; open, non-proprietary data formats; clear, consistent meta-data, using international standards for data structure where available; and licensed for re-use through CC BY). To balance the needs of trial participants for protection of their sensitive health data (in accordance with informed consent) and the needs of the scientific community for data availability, we will follow the principle "as closed as necessary, as open as possible". Results summaries will also be posted at Clinicaltrials.gov after the project end.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of summary results; no end date
Access Criteria: Openly accessible